CLINICAL TRIAL: NCT02889783
Title: Urethral Sensory Profile: a New Technique to Evaluate Urethral Sensation Prospective Evaluation in Patients With or Without Neurological Disorders
Status: Completed | Type: Observational
Sponsor: Groupe de Recherche Clinique en Neuro-Urologie (Other)
Responsible Party: Principal Investigator, Amarenco, Gerard Amarenco, MD PHD, Groupe de Recherche Clinique en Neuro-Urologie
Other Study IDs: GREEN-1-LW
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Urethral Cyst
Keywords: urodynamics; urethral sensation; urethral pain

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: record of urethral pain sensation during urodynamics study — Record of pain using a VAS scale during the first catheterizing of urodynamics study, at every centimeter

SUMMARY:
This is a routine evaluation of urethral sensation during urodynamic studies. The record has been realized retrospectively. The investigators propose a new way to represent urethral sensation, in a simple and non-invasive way.

DETAILED DESCRIPTION:
All patients consulting for urodynamics were included. During the introduction of the urinary catheter for urodynamic evaluation, patients were asked to report pain and/or desire to void felt at every centimeter (cm)of insertion, on an analogic visual scale graded from 0 to 10. The USP was defined by the graphic representation of the successive values of these sensations , from the urinary meatus, to the urinary bladder.

ELIGIBILITY:
Inclusion Criteria:

* patients consulting in our department for a urodynamic study

Exclusion Criteria:

* chronic pelvic pain
* difficulties for understanding or for communicating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients consulting for an urodynamic study in our tertiary care unit.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Urethral Sensitive profile | mars 2015
  record of urethral pain sensation during the first catheterizing of urodynamics study

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Amarenco, MD PHD, Principal Investigator — UPMC, Sorbonne Université, Univ Paris 6, service neuro-urologie, hôpital TENON, Paris
Locations (1):
- Weglinski, Paris, France

IPD SHARING:
Plan to Share IPD: No